CLINICAL TRIAL: NCT04474158
Title: Creating Peace: Community-based Youth Violence Prevention to Address Racism and Discrimination
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Elizabeth Miller, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY18110082; 5R01MD013797-02 (NIH)
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Adolescent Behavior; Group, Peer; Violence, Non-accidental; Violence, Sexual; Violence, Domestic; Emotional Abuse; Coping Skills; Communication, Personal
MeSH Terms: conditions — Adolescent Behavior; Coitus; Communication

STUDY DESIGN:
Intervention Model Description: This cluster-randomized community-partnered study will examine the effectiveness of a trauma-sensitive, gender transformative youth violence prevention program called Creating Peace that integrates racism and discrimination prevention among youth ages 14-19. The study will be located in Pittsburgh, Pennsylvania across 24 neighborhoods with concentrated disadvantage ('clusters'), randomized either to receive the "Creating Peace" program (i.e., intervention neighborhood, n=12) or to a job skills training program (n=12 schools).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creating Peace (Experimental): Creating Peace uses a group discussion format with activities that explore race, gender, sexual identity, and social class. Creating Peace is a 12 session curriculum designed to support youth ages 14-19 in healing from experiences of trauma by restoring social connections, strengthening positive coping strategies that exclude all forms of violence, challenging gender norms that foster violence perpetration, and practicing positive bystander intervention skills to intervene safely with peers' disrespectful and harmful behaviors. Through 12 sessions (3 hours/session) over a 4 to 12 week period, Creating Peace offers gender transformative content combined with youth leadership development. Near program conclusion, youth will offer guidance to law enforcement on interacting with youth in a process of social restoration.
  Interventions: Behavioral: Creating Peace
- Job Readiness Training (Active Comparator): Job Readiness Training uses a group discussion format to learn specific skills to prepare for employment including developing goals, seeking jobs, preparing for interviews, and so forth. Participants receive a 12 session job readiness training with linkages to businesses and employment opportunities. Discussions include a wide range of topics related to career exploration and job readiness.
  Interventions: Behavioral: Job Readiness

INTERVENTIONS:
Behavioral: Creating Peace — Creating Peace is a 12 session curriculum designed to support youth ages 14-19 in healing from experiences of trauma by restoring social connections, strengthening positive coping strategies that exclude all forms of violence, challenging gender norms that foster violence perpetration, and practicing positive bystander intervention skills to intervene safely with peers' disrespectful and harmful behaviors. Through 12 sessions (3 hours/session) over a 4 to 12 week period, Creating Peace offers gender transformative content combined with youth leadership development. Near program conclusion, youth will offer guidance to law enforcement on interacting with youth in a process of social restoration.
  Arms: Creating Peace
Behavioral: Job Readiness — Job Readiness Training uses a group discussion format to learn specific skills to prepare for employment including developing goals, seeking jobs, preparing for interviews, and so forth.
  Arms: Job Readiness Training

SUMMARY:
This cluster-randomized community-partnered study will examine the effectiveness of a trauma-sensitive, gender transformative youth violence prevention program called Creating Peace that integrates racism and discrimination prevention with youth ages 14-19.

DETAILED DESCRIPTION:
This community-partnered cluster-randomized controlled trial will examine the effectiveness of a trauma-sensitive, gender-transformative youth violence prevention program that integrates racism and discrimination prevention.

Set in 24 neighborhoods in Pittsburgh, Pennsylvania with concentrated social and economic disadvantage, this study addresses gender and racial injustice through a series of group discussions, bringing together adolescents ages 14-19 with law enforcement officers in a process of social restoration.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ages 14-19 (inclusive)
* Participants must speak English

Exclusion Criteria:

* Not ages 14-19 (inclusive)
* Do not speak English

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participants that self report any self-representation of gender identity to include, but not limited to, male, female, trans-male, trans-female or gender non conforming.
Enrollment: 1800 (Estimated)
Dates: Start 2020-12-04 (Actual); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-02-23 (Estimated)

PRIMARY OUTCOMES:
Change in recent use of any violence at 3 months | At baseline and three months after program conclusion
  Summary score of any recent use of violence (physical, sexual, and emotional abuse; sexual violence; physical violence and threatening with a weapon; cyber dating abuse, cyber peer abuse, and sexting) calculated as one point for each behavior then summed (lower score indicates better outcome)
Change in recent use of any violence at 9 months | At baseline and nine months after program.
  Summary score of any recent use of violence (physical, sexual, and emotional abuse; sexual violence; physical violence and threatening with a weapon; cyber dating abuse, cyber peer abuse, and sexting) calculated as one point for each behavior then summed (lower score indicates better outcome)

SECONDARY OUTCOMES:
Change in past 30 day weapon carrying at 3 months | At baseline and three months after program conclusion
  Self-reported number of days they carried a weapon in past 30 days
Change in past 30 day weapon carrying at 9 months | At baseline and nine months after program conclusion
  Self-reported number of days they carried a weapon in past 30 days
Change in positive bystander behaviors at 3 months | At baseline and three months after program conclusion
  Past 3 month positive bystander behavior when witnessing disrespectful and harmful behavior among peers comparing baseline and follow up summary scores. Participants report if they have witnessed peers' abusive behaviors in the past 3 months and if witnessed, how they responded (whether they intervened to interrupt the behavior, provided support to person being harmed).
Change in positive bystander behaviors at 9 months | At baseline and nine months after program conclusion
  Past 3 month positive bystander behavior when witnessing disrespectful and harmful behavior among peers comparing baseline and follow up summary scores. Participants report if they have witnessed peers' abusive behaviors in the past 3 months and if witnessed, how they responded (whether they intervened to interrupt the behavior, provided support to person being harmed).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The research team will not make individual participant data (IPD) available to other researchers.